CLINICAL TRIAL: NCT03740750
Title: The Effect of 4 Hours of Tens and Heat on Pain and Range of Motion in the Lower Back and the Duration of Pain Relief After Tens and Heat Are Removed
Brief Title: TENS and Heat for Reducing Back Pain in Humans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Future Sciene Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: jand m18
Record Dates: First submitted 2018-11-08; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Pain
Keywords: heat; hot temperature; cutaneous electrostimulation
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: 6 different interventions will be tested in parallel on 6 equivalent groups of subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- control (Placebo Comparator): sham heat and sham TENS
  Interventions: Device: sham heat; Device: sham Tens
- heat only (Experimental): heat applied to the back for 4 hours with sham TENS
  Interventions: Device: Thermacare heat wraps; Device: sham Tens
- Tens only (Experimental): Tens applied for 4 hours with sham heat
  Interventions: Device: TENS; Device: sham heat
- Heat and Tens continuous (Experimental): Heat and Tens applied together for 4 hours
  Interventions: Device: Thermacare heat wraps; Device: TENS
- Tens 15 (Experimental): Tens applied only 15 minutes each hour for 4 hours, sham heat
  Interventions: Device: TENS; Device: sham heat
- Heat and Tens 15 (Experimental): Heat applied for 4 hours with tens only applied the last 15 minutes of each hour
  Interventions: Device: Thermacare heat wraps; Device: TENS

INTERVENTIONS:
Device: Thermacare heat wraps — low level continuous heat wrap
  Arms: Heat and Tens 15; Heat and Tens continuous; heat only
Device: TENS — electrical stimulation
  Arms: Heat and Tens 15; Heat and Tens continuous; Tens 15; Tens only
Device: sham heat — expended heat wrap
  Arms: Tens 15; Tens only; control
Device: sham Tens — tens applied but unit not turned on
  Arms: control; heat only

SUMMARY:
Lower back pain is one of the most common and most expensive impairments costing time and expense in the work force today. With the effects on cognitive skills and addictive side effects of opioids and other prescription pain killers, there has been increasing interest in alternative medical treatments to relieve pain. Two of these that are commonly used are heat and transcutaneous electrical nerve stimulation (TENS). In the present investigation, there are two objectives 1) to determine if Tens needs to be continuous or can be intermittent and still achieve pain relief and 2) To see how long pain relief lasts after 4 hours of application of tens, heat or both. There will be seventy-five subjects with chronic back pain divided into 6 groups randomly; 15 subjects per group. The intervention will be either TENS alone, Heat alone or Tens plus heat or a control group.

DETAILED DESCRIPTION:
There will be seventy-five subjects with chronic back pain divided into 6 groups randomly; 15 subjects per group. They are between the ages of 24 and 60 years old. They will not be taking pain medications for at least 48 hours prior to the study. The groups were as follows;

1. Control
2. heat only
3. Tens only
4. Tens and heat
5. Tens for the last 15 minutes each hour plus heat
6. Tens for the last 15 minutes each hour Tens is at threshold intensity (12 ma) at a frequency of 20 Hz either ramped continuously or for the last 15 minutes of each hour. The stimulation is 3 seconds increase to threshold, 3 seconds hold and 3 seconds ramped down followed by a 9 second rest period. Pain is assessed by an analog visual pain scale and an algometer placing pressure on the back to assess the pressure that causes pain, a measure of inflammation. In addition, the Oswestry lower back pain index and Roland Morris questionnaire are used. Range of motion in the trunk where first pain is felt is also measured.

ELIGIBILITY:
Inclusion Criteria:

1. pain for at least 3 months in the lower back
2. age range 24-60

Exclusion Criteria:

1. Those with back pain caused by fractures or spinal damage
2. those who had undergone low back surgery within the last year
3. those with diagnosed diabetes
4. no use of opiod pain meds for at least 10 days

Ages: 24 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
range of motion of the hip for flexion, extension,left and right rotation,left and right bending | Baseline (beginning of study before intervention)
  range of motion in 6 degrees of freedom in the lower back
subjective pain by marking on scale | Baseline (beginning of study before intervention)
  analog visual pain scale on separate piece of paper 10cm in length- subject marks pain level with 10 the worst
pressure on back that causes pain | Baseline (beginning of study before intervention)
  pressure applied to lower back until pain is felt to assess inflammation
range of motion of the hip for flexion, extension,left and right rotation,left and right bending | 4 hours after study start- at end of intervention
  range of motion in 6 degrees of freedom in the lower back
subjective pain by marking on scale | 4 hours after study start- at end of intervention
  analog visual pain scale on separate piece of paper 10cm in length- subject marks pain level with 10 the worst
pressure on back that causes pain | 4 hours after study start- at end of intervention
  pressure applied to lower back until pain is felt to assess inflammation
range of motion of the hip for flexion, extension,left and right rotation,left and right bending | 10 hours after study start( 6 hours after the modality ends)
  range of motion in 6 degrees of freedom in the lower back
subjective pain by marking on scale | 10 hours after study start( 6 hours after the modality ends)
  analog visual pain scale on separate piece of paper 10cm in length- subject marks pain level with 10 the worst
pressure on back that causes pain | 10 hours after study start( 6 hours after the modality ends)
  pressure applied to lower back until pain is felt to assess inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Mike Laymon, PT, DSC, Study Director — Future Science Technology
Locations (1):
- Future Sciecne Technology, Henderson, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Petrofsky J, Laymon M, Khowailed I, Lee H. Synergistic Effects of Continuous Low Level Heat Wraps and Vitamins in Improving Balance and Gait in Adults. Int J Vitam Nutr Res. 2016 Jun;86(3-4):152-160. doi: 10.1024/0300-9831/a000428. Epub 2018 Jan 30. PMID 29381114
- [Result] Petrofsky JS, Laymon M, Alshammari F, Khowailed IA, Lee H. Use of low level of continuous heat and Ibuprofen as an adjunct to physical therapy improves pain relief, range of motion and the compliance for home exercise in patients with nonspecific neck pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2017;30(4):889-896. doi: 10.3233/BMR-160577. PMID 28282796
- [Result] Stark J, Petrofsky J, Berk L, Bains G, Chen S, Doyle G. Continuous low-level heatwrap therapy relieves low back pain and reduces muscle stiffness. Phys Sportsmed. 2014 Nov;42(4):39-48. doi: 10.3810/psm.2014.11.2090. PMID 25419887